CLINICAL TRIAL: NCT01058252
Title: A Scientific & Clinical Review of Minimal Stimulation Protocol Using AROMEK (Letrozole) and Follitrope (Recombinant FSH)Combined With INVOCell(Intravaginal Culturing) - Effectiveness as Low Cost IVF
Brief Title: Minimal Stimulation Protocol Using Aromek(Letrozole) and Follitrope(recFSH) Combined With INVOCell-Low Cost IVF
Acronym: MSP-INVO IVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Galaxy Pharma (Pvt) Limited (Industry)
Collaborators: Ova IVF & Reproductive Health Clinics, Karachi (Unknown)
Responsible Party: Sponsor
Other Study IDs: GIVF-SRM 1001
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Primary Infertility; Secondary Infertility; Low Responders; Mild to Moderate Male Factor Infertility
MeSH Terms: interventions — Letrozole; Indomethacin; Embryo Transfer; Contraceptive Devices, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Letrozole, recFSH, INVOCell, Monitoring: Infertile couple following MSP with INVO IVF
  Interventions: Combination Product: INVOCell, Letrozole 2.5 mg, recFSH 75 IU; Procedure: STEP-3: LH Suppression & Monitoring; Procedure: STEP-4: HCG Timing; Procedure: STEP-5: OPU, ET, Cancellation; Procedure: INVOCell (Intravaginal Culturing)

INTERVENTIONS:
Combination Product: INVOCell, Letrozole 2.5 mg, recFSH 75 IU — OVARIAN STIMULATION:
  In previous cycles, cycle length and ovulatory status must be assessed and documented.
  STEP 1: ANOVULATION by ORAL CONTRACEPTION
  * Place patients on monophasic low dose of oral contraceptive pills (OCP) such as Marvelon (Organon, 0.03 mg) continuously for 21 days, 22 days but no more.
  * Before stopping the oral contraceptive pills, perform an ultrasound to check for the absence of cysts (no cyst > 10 mm).
  * Give estradiol (2mg, 3 times a day) for 3 days from D21 or D22 and wait for bleeding.
  STEP 2: STIMULATION and MONITORING Day one of the cycle equals the first day of bleeding (not spotting).
  * On Day 3 (D3), start letrozol 2.5mg (AROMEK) for 5 days (D7). LetrozolE can be pushed for 2 more days.
  * Start hMG or FSH (75 IU a day) on Day 3 like LetrozolE and continue for 5 to 7 days without increasing the dose. The dose of hMG OR FSH can be increased to 150 IU a day if low responder.
  Other Names: Aromek (Letrozole 2.5 mg);; Follitrope (Recombinent FSH - 75 IU); IVF-C 5000 IU (HCG); Ova-Surge (Urinary LH Surge Kit); Indomethacin 50 mg
Procedure: STEP-3: LH Suppression & Monitoring — Baseline Day-2 Ultrasound to estimate antral follicles; Follow-up TVS scans on Day- 5,6,7,8 and 9 of the stimulated cycle. Ideally the lead follicle should be 18 mm on or around day 10 of the cycle.
  • When the leading follicle reaches 14 to15 mm (D8 or D9), give Indomethacine (50 mg, 3 times a day) until the evening preceding the egg retrieval. The Indomethacine will prevent a premature ovulation.
  The endometrium should be minimum 8 mm on the day of HCG (IVF-C 5000 IU x 2)
  No need of LH testing, or E2 testsing during the stimulated cycle.
Procedure: STEP-4: HCG Timing — IVF-C (HCG 10000 IU) shall be injected to trigger the ovulation, when any of the following occur:
  * E2 level is over 150 pg/ml/per mature follicle (> 15 mm)
  * Domminent follicle is greater than 18 mm in mean diameter
  * LH Remains as Baseline, OR
  * The day when Urinary LH Surge is positive
  Other Names: IVF-C 5000 IU
Procedure: STEP-5: OPU, ET, Cancellation — Ultrasound guided Ovum Pick-Up is performed 34-36 hours after IVF-C (HCG 10000 IU) injection.
  Embryo Transfer is performed after 48-72 hours of incubation at 4-8 cell stage.
  Maximum of 2 embryos are transferred, using ultrasound guided transfer.
  Cancellation Criteria:
  * Poor patient compliance
  * Premature Ovulation
  * Premature LH Surge
  * Endometrium < 7 mm
  * Poor Follicular Development
  * E2 Level > 2,500 pg/ml
  Other Names: Ovum Pick-Up; Embryo Transfer; Ultrasound Guided
Procedure: INVOCell (Intravaginal Culturing) — Sperm preparation through Swim-Up or Gradient is performed 1 hour prior to the oocyte retrieval; Fill the device without air bubble. Only 100000 motile spermatozoa are added into the device; After follicle aspiration, oocyte(s) are identified in the follicular fluid and immediately placed into the device; The device is closed, placed into a protective outer rigid shell and then positioned into the vaginal cavity for 2 to 3 days; No activity restriction is required for the patient, except baths. After 2 or 3 days of incubation, the retention system and the device are removed from the vagina in sterile environment. The device is opened and the contents are observed in a sterile environment under microscope to find the embryos. The two best quality embryos are loaded into embryo transfer catheter and transferred immediately unto the uterine cavity using aseptic techniques.
  Other Names: INVOCell; Diaphragm (Retention Device)

SUMMARY:
The purpose of this study to evaluate a low cost minimal stimulation protocol combined with Intravaginal Culturing, to make IVF affordable and available across the large infertile/subfertile population

DETAILED DESCRIPTION:
In routine ART procedures for IVF, ovarian stimulation is performed using down regulation with GNRH Agonist combined with high daily FSH doses followed with ovulation induction with HCG 10000 IU, ovum pick-up 34-36 hours after HCG injection and embryo transfer on day 2, 3 or 5.

In routine ART procedure for IVF, embryology is done in very high tech lab, contamination free environment, which also exclude VOC, high quality CO2 Incubators, laminar flow with heated table top, high magnification stereo microscope along with equipments for maintaining quality control, with a highly trained embryologist. The primary reason is we need to create a womb like environment in the embryology lab as eggs, and mainly fertilised embryos are going to spend minimum 2 or 3 and in case blastocyst 5 days in this lab.

In recent years, various studies have been published identifying various minimal stimulation protocols for IVF, and also another variation of IVF where rather than using CO2 Incubator for culturing, vaginal cavity of the female partner is used for incubation using a specially designed capsule which have walls permeable to vaginal pCO2 and O2. Oocytes are retrieved by the physician and handed over to basic embryologist to identify and grade oocytes and washed sperms are placed in a embryo toxic tested, sterile, individual single use capsule (INVOCell) and placed in vaginal cavity using diaphragm, patient goes back to home with some instructions for care, on day 2 patient comes back to the IVF Clinic and physician gets the capsule out and hands over to the basic embryologist trained on INVOCell to identify embryos and grade them, further loading of embryos on ET Catheter.

ELIGIBILITY:
Inclusion Criteria:

* Tubal factor without Hydrosalpinx
* Unexplained infertility with unsuccessful attempts in achieving pregnancy through timed intercourse or IUI
* Boarder line male factor infertility
* Sperm DNA Fragmentation < 30%
* Normal Uterine Cavity
* Normal baseline ultrasound with adequate number of primary follicles present
* Normal FSH and E2 on Day 3
* Age of the female is < 35 years old

Exclusion Criteria:

* If previous IVF or INVO attempts resulted in failed fertilisation
* Male partner who has difficulty in producing semen sample
* Very low sperm count, very low percentage of sperm motility and morphology
* Sperm DNA Fragmentation > 30%
* Age of female patient > 37 years
* Borderline or elevated E2 or FSH on day 3 or failed CCCT or low blood inhibin levels
* Poor ovarian response
* Hydrosalpinx
* Anatomic difficulties in reaching ovaries for oocyte retrieval
* Cervical stenosis, making embryo transfer difficult
* Uterine abnormalities or deformities
* Obesity

Ages: 20 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: IVF Network Centers across the country, selecting patients meeting inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Number of Follicles >18 mm on the day of HCG; Number of Oocytes aspirated; Fertilisation Rate | Quarterly

SECONDARY OUTCOMES:
Pregnancy Rate; Cost of Treatment | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gul Rana, MBBS, Study Director — Ova IVF & Reproductive Health Clinics
Locations (2):
- Pakistan (2):
  - Lady Wallington Hospital, Lahore, Punjab Province
  - Ova IVF & Reproductive Health Clinics, Karachi, Sindh

REFERENCES:
- [Background] Hewitt J. Intravaginal culture: present and potential uses. Br J Hosp Med. 1990 Sep;44(3):182, 184-5, 188. PMID 2257400
- [Result] Ranoux C, Poirot C, Foulot H, Aubriot FX, Dubuisson JB, Chevallier O. [Intravaginal culture and embryo transfer]. Rev Fr Gynecol Obstet. 1988 Oct;83(10):637-8. French. PMID 3201055
- [Result] Ranoux C, Aubriot FX, Dubuisson JB, Cardone V, Foulot H, Poirot C, Chevallier O. A new in vitro fertilization technique: intravaginal culture. Fertil Steril. 1988 Apr;49(4):654-7. doi: 10.1016/s0015-0282(16)59835-5. PMID 3350160
- [Result] Sterzik K, Rosenbusch B, Sasse V, Wolf A, Beier HM, Lauritzen C. A new variation of in-vitro fertilization: intravaginal culture of human oocytes and cleavage stages. Hum Reprod. 1989 Nov;4(8 Suppl):83-6. doi: 10.1093/humrep/4.suppl_1.83. PMID 2613877
- [Result] Freude G, Artner B, Leodolter S. [Intravaginal culture--simplification of IVF]. Wien Med Wochenschr. 1990 Oct 31;140(20):498-501. German. PMID 2264352
- [Result] Sterzik K, Rosenbusch B, Sasse V, Terinde R, Wolf A, Beier HM, Lauritzen C. [Experiences and successes with intravaginal fertilization and culture of human oocytes]. Geburtshilfe Frauenheilkd. 1988 Dec;48(12):850-3. doi: 10.1055/s-2008-1026639. German. PMID 3234716
- [Result] Sh Tehrani Nejad E, Abediasl Z, Rashidi BH, Azimi Nekoo E, Shariat M, Amirchaghmaghi E. Comparison of the efficacy of the aromatase inhibitor letrozole and clomiphen citrate gonadotropins in controlled ovarian hyperstimulation: a prospective, simply randomized, clinical trial. J Assist Reprod Genet. 2008 May;25(5):187-90. doi: 10.1007/s10815-008-9209-2. Epub 2008 Apr 19. PMID 18427974
- [Result] Grabia A, Papier S, Pesce R, Mlayes L, Kopelman S, Sueldo C. Preliminary experience with a low-cost stimulation protocol that includes letrozole and human menopausal gonadotropins in normal responders for assisted reproductive technologies. Fertil Steril. 2006 Oct;86(4):1026-8. doi: 10.1016/j.fertnstert.2006.03.034. Epub 2006 Aug 28. PMID 16935285
- [Result] Baysoy A, Serdaroglu H, Jamal H, Karatekeli E, Ozornek H, Attar E. Letrozole versus human menopausal gonadotrophin in women undergoing intrauterine insemination. Reprod Biomed Online. 2006 Aug;13(2):208-12. doi: 10.1016/s1472-6483(10)60617-7. PMID 16895634
- [Result] Jee BC, Ku SY, Suh CS, Kim KC, Lee WD, Kim SH. Use of letrozole versus clomiphene citrate combined with gonadotropins in intrauterine insemination cycles: a pilot study. Fertil Steril. 2006 Jun;85(6):1774-7. doi: 10.1016/j.fertnstert.2006.02.070. Epub 2006 May 4. PMID 16677640
- [Result] Garcia-Velasco JA, Moreno L, Pacheco A, Guillen A, Duque L, Requena A, Pellicer A. The aromatase inhibitor letrozole increases the concentration of intraovarian androgens and improves in vitro fertilization outcome in low responder patients: a pilot study. Fertil Steril. 2005 Jul;84(1):82-7. doi: 10.1016/j.fertnstert.2005.01.117. PMID 16009161
- [Result] Verpoest WM, Kolibianakis E, Papanikolaou E, Smitz J, Van Steirteghem A, Devroey P. Aromatase inhibitors in ovarian stimulation for IVF/ICSI: a pilot study. Reprod Biomed Online. 2006 Aug;13(2):166-72. doi: 10.1016/s1472-6483(10)60611-6. PMID 16895628
- [Result] Ozmen B, Sonmezer M, Atabekoglu CS, Olmus H. Use of aromatase inhibitors in poor-responder patients receiving GnRH antagonist protocols. Reprod Biomed Online. 2009 Oct;19(4):478-85. doi: 10.1016/j.rbmo.2009.05.007. PMID 19909587
- [Result] Goswami SK, Das T, Chattopadhyay R, Sawhney V, Kumar J, Chaudhury K, Chakravarty BN, Kabir SN. A randomized single-blind controlled trial of letrozole as a low-cost IVF protocol in women with poor ovarian response: a preliminary report. Hum Reprod. 2004 Sep;19(9):2031-5. doi: 10.1093/humrep/deh359. Epub 2004 Jun 24. PMID 15217999
- [Result] Kadoch IJ, Al-Khaduri M, Phillips SJ, Lapensee L, Couturier B, Hemmings R, Bissonnette F. Spontaneous ovulation rate before oocyte retrieval in modified natural cycle IVF with and without indomethacin. Reprod Biomed Online. 2008 Feb;16(2):245-9. doi: 10.1016/s1472-6483(10)60581-0. PMID 18284881
- [Result] Janssens RM, Lambalk CB, Vermeiden JP, Schats R, Schoemaker J. In-vitro fertilization in a spontaneous cycle: easy, cheap and realistic. Hum Reprod. 2000 Feb;15(2):314-8. doi: 10.1093/humrep/15.2.314. PMID 10655301
- [Result] Bernabeu R, Roca M, Torres A, Ten J. Indomethacin effect on implantation rates in oocyte recipients. Hum Reprod. 2006 Feb;21(2):364-9. doi: 10.1093/humrep/dei343. Epub 2005 Nov 10. PMID 16284067
- [Result] Khan M, Zafar S, Syed S. Successful intravaginal culture of human embryos for the first time in Pakistan--an experience at the Sindh Institute of Reproductive Medicine, Karachi. J Pak Med Assoc. 2013 May;63(5):630-2. PMID 23757995
- [Result] Lucena E, Saa AM, Navarro DE, Pulido C, Lombana O, Moran A. INVO procedure: minimally invasive IVF as an alternative treatment option for infertile couples. ScientificWorldJournal. 2012;2012:571596. doi: 10.1100/2012/571596. Epub 2012 May 2. PMID 22645435
- [Result] Doody KJ, Broome EJ, Doody KM. Comparing blastocyst quality and live birth rates of intravaginal culture using INVOcell to traditional in vitro incubation in a randomized open-label prospective controlled trial. J Assist Reprod Genet. 2016 Apr;33(4):495-500. doi: 10.1007/s10815-016-0661-0. Epub 2016 Feb 3. PMID 26843390
- [Result] Babcock Gilbert S, Polotsky AJ. Vaginal culture for IVF allows two mothers to carry the same pregnancy: Is more always better? Case Rep Womens Health. 2019 Jan 26;21:e00099. doi: 10.1016/j.crwh.2019.e00099. eCollection 2019 Jan. PMID 30733926
- [Result] Garcia-Ferreyra J, Hilario R, Luna D, Villegas L, Romero R, Zavala P, Duenas-Chacon J. In Vivo Culture System Using the INVOcell Device Shows Similar Pregnancy and Implantation Rates to Those Obtained from In Vivo Culture System in ICSI Procedures. Clin Med Insights Reprod Health. 2015 Jun 10;9:7-11. doi: 10.4137/CMRH.S25494. eCollection 2015. PMID 26085790
- [Result] Mitri F, Esfandiari N, Coogan-Prewer J, Chang P, Bentov Y, McNaught J, Klement AH, Casper RF. A pilot study to evaluate a device for the intravaginal culture of embryos. Reprod Biomed Online. 2015 Dec;31(6):732-8. doi: 10.1016/j.rbmo.2015.09.005. Epub 2015 Sep 18. PMID 26602106
- See also: Real-world experience with intravaginal culture using INVOCELL: an alternative model for infertility treatment — https://www.researchgate.net/publication/347083270_Real-world_experience_with_intravaginal_culture_using_INVOCELL_an_alternative_model_for_infertility_treatment